CLINICAL TRIAL: NCT06220019
Title: REspiratory diSEAse cohoRt Studies of CHinese Medicine for Pneumonia (RESEARCH-Pneumonia)
Status: Not yet recruiting | Type: Observational
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Wuhan No.1 Hospital (Other); Hebei Provincial Hospital of Traditional Chinese Medicine (Other Government); Shanghai University of Traditional Chinese Medicine (Other); Qingdao Hiser Medical Group (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Shaanxi Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RESEARCH-Pneumonia
Record Dates: First submitted 2024-01-05; First posted 2024-01-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-09

CONDITIONS: Pneumonia
Keywords: Pneumonia; Chinese Medicine; Cohort
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The biological sample bank includes serum samples, plasma samples, urine samples, stool samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TCM Group: The study will include adult patients discharged after hospitalization for pneumonia, with no restrictions on TCM syndromes. Patients diagnosed with pneumonia via laboratory or imaging tests at admission and treated in the hospital will be eligible if enrolled within seven days of discharge. Follow-ups will occur every three months over one year, documenting treatment methods (TCM or Western medicine), hospitalizations, respiratory infections, mortality, and quality of life.
  Subgroup analyses will be conducted based on age, type of pneumonia (community- or hospital-acquired), specific TCM treatments (e.g., Chinese patent medicines or external therapies), and treatment duration.
  Interventions: Drug: TCM
- Non-TCM Group: All patients who do not meet the defined criteria for the TCM group will be classified into the non-TCM group.

INTERVENTIONS:
Drug: TCM — We will perform subgroup analyses based on specific TCM interventions (such as Chinese patent medicines or external therapies) and the duration of TCM treatment (for example, comparing patients who receive continuous oral Chinese patent medicine for two months or more each year with those who do not). These analyses will assess the efficacy and safety of TCM.
  Groups: TCM Group

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of dialectical treatment in the patients with pneumonia after discharge in a prospective cohort study: one is the Traditional Chinese Medicine (TCM) cohort, which has been evaluated and has certain effects; The other is a non traditional Chinese medicine queue.

DETAILED DESCRIPTION:
The incidence, hospitalization rate, and mortality associated with pneumonia are significant, contributing to a substantial disease burden. Post-discharge follow-up and intervention strategies for pneumonia patients are often insufficient, leaving patients vulnerable to readmission or mortality due to recurrent pneumonia and related complications. In clinical practice, there is a predominant focus on the amelioration of clinical symptoms during hospitalization, with limited attention to ongoing outpatient interventions aimed at reducing readmission rates. Consequently, there is a pressing need for cohort studies on pneumonia.

This study is a multicenter, prospective cohort study involving adult patients discharged after pneumonia treatment. Approximately 5,000 patients will be enrolled, with follow-up assessments conducted every three months over the course of one year. After one year, patients will be stratified into two cohorts based on the duration of Traditional Chinese medicine (TCM) treatment received (e.g., continuous treatment for two months or intermittent treatment for three months per year). One cohort will consist of patients receiving TCM, while the other will include those who did not receive TCM. The primary endpoint is the rate of hospital readmission, while secondary outcomes include treatment satisfaction, physician-reported outcomes, patient-reported outcomes, quality of life, nutritional status, incidence of acute upper respiratory tract infections, and survival. This study aims to evaluate the clinical efficacy and safety of TCM in the management of adult pneumonia patients following discharge.

ELIGIBILITY:
Selection Criteria:

* Hospitalized patients with a confirmed diagnosis of pneumonia (HAP, CAP).
* Age ≥18 years.
* Signed informed consent form.

Exclusion Criteria:

* Patients with confusion, consciousness disorders, dementia, and various mental illnesses;
* Patients with altered mental status, dementia, consciousness disorders, or various psychiatric conditions;
* Those who are completely unable to care for themselves or are bedridden long-term; and those currently participating in other clinical drug trials.
* Known to be allergic to treatment drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients discharged after pneumonia.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization rate | The Rehospitalization rate within a one-year follow-up period
  Including all-cause readmission rate and pulmonary infection readmission rate

SECONDARY OUTCOMES:
Patient satisfaction with efficacy | Changes in ESQ-COPD relative to baseline at months 3, 6, 9, and 12 during the follow-up phase
  The Effectiveness Satisfaction Questionnaire of CAP (ESQ-CAP) was used to evaluate the efficacy of pneumonia patients.
Health survey summary table（SF-36） | Changes in SF-36 relative to baseline at months 3, 6, 9, and 12 during the follow-up phase
  Using SF-36 to evaluate the impact of CAP on a person's life over time
Clinical outcomes reported by patients | Changes in CAP-PRO relative to baseline at months 3, 6, 9, and 12 during the follow-up phase
  The Patient Reported Outcome for CAP (CAP-PRO) was used to assess the quality of life and health status of patients with pneumonia.
Clinical outcomes reported by doctors | Changes in CAP-CRO relative to baseline at months 3, 6, 9, and 12 during the follow-up phase
  The Clinical Reported Outcome for CAP (CAP CRO) was used to assess the patient's condition.
nutritional status | Changes in nutritional status of CAP patients relative to baseline at 6 and 12 months of follow-up stage
  Nutritional status related indicators.
Acute upper respiratory tract infection (URTI) event | Acute upper respiratory tract infection events that occurred during the one-year follow-up period
  It is a general term for acute inflammation of the nose, pharynx, or throat caused by various viruses and/or bacteria, including common cold, acute viral pharyngitis or laryngitis, acute herpetic pharyngitis, pharyngoconjunctival fever, bacterial pharyngitis, and tonsillitis.
Survival situation | Changes in patient survival situation relative to baseline at months 3, 6, 9, and 12 during the follow-up phase
  Record the number of deaths. Record the follow-up period every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, Doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No